CLINICAL TRIAL: NCT04697095
Title: Survival of Monocytes Collected From Patients With Atrophic AMD in Retinal Pigmented Epithelium Explants
Acronym: SURViVOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL20_0027
Record Dates: First submitted 2020-12-22; First posted 2021-01-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration
Keywords: Wet AMD; Dry AMD; Monocytes; Survival; Cytokines; Inflammation; Blood Samples
MeSH Terms: conditions — Macular Degeneration; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- early / intermediate AMD without neovessels and without macular atrophy (Experimental)
  Interventions: Other: Blood samples
- Late exsudative AMD with neovessels (Experimental)
  Interventions: Other: Blood samples
- Late AMD with macular atrophy without neovessels (Experimental)
  Interventions: Other: Blood samples
- Patientes with No AMD (Sham Comparator)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — : The blood sample from all groups will be taken on the day of inclusion, in the ophthalmology department. The patient will be cared for by a nurse and then taken to the collection room. A 100 ml sample will be taken (10 tubes of 10 ml). Blood samples will be labeled with the patient's identification number as part of the protocol. They will be transported to the research laboratory in order to be picked up for monocyte extraction. The purification of blood monocytes will be done. In case of excess, the samples will be destroyed at the end of the study.

SUMMARY:
Age-related macular degeneration (AMD) affects 2 million people in France and is the main cause of irreversible blindness in France. All patients initially have an early form of the disease. This early form can evolve in two different ways: the atrophic form, which progresses slowly, and the exudative or neovascular form, which has a more rapid evolution. While there are treatments for the exudative form of the disease, there is currently no therapy for the atrophic form of AMD. Recently, it has been demonstrated in atrophic AMD that there is accumulation of inflammatory cells, monocytes, in the sub-retinal space. This space is located between the retinal pigment epithelium (RPE) and photoreceptors. It is physiologically devoid of immune cells (immune privilege). Monocytes secrete many pro-inflammatory molecules, such as cytokines. Some cytokines (IL-1, IL6 and TNF) have a deleterious role on RPE and photoreceptors in mouse models. The identification of specific cytokines would help to better understand this disease and consider potential targeted therapies. Our project is based on the hypothesis that monocytes extracted from patients with AMD have a superior survival on RPE compared to monocytes extracted from healthy patients (without retinal pathology), and more particularly in atrophic forms of AMD. The main aim of this study is to compare the survival of monocytes extracted from patients with atrophic AMD to monocytes extracted from patients without retinal pathology (control) on retinal pigment epithelial cell lines (ARPE-19). Survival will be evaluated by automated counting of monocytes after 24 hours of culture on ARPE-19 after specific immunostaining of monocytes. If the survival of monocytes from patients with the late form of AMD is increased then therapy directly targeting this pathological accumulation of monocytes could be considered. Moreover, the identification of increased secretion of certain cytokines and the demonstration of their deleterious effect on retinal physiology could lead to targeted therapies against them.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Male or female older than 50,
* Provide written informed consent,
* Patient affiliated to French social security,
* Maximum sampling volume (care + research) per 30-day period to be adapted according to the weight of the patient

Specific criteria:

Patient presenting in both eyes:

* Either the same type of AMD defined according to the modified international AREDS study (Ferris et al. 2013),
* or early AMD in one eye and atrophic AMD in the other eye, the patient will therefore be defined as being atrophic
* or early AMD in one eye and exudative AMD in the other eye, the patient will therefore be defined as exudative,
* or no retinal pathology (control group).

Exclusion Criteria:

General criteria:

* Patient whose weight is less than 50kg,
* Adult patient under guardianship or curatorship or unable to express consent,
* Person deprived of liberty,
* Patient participating in an ongoing clinical trial during the inclusion visit,

Specific criteria:

* Patient with atrophic AMD in one eye and exudative AMD in the other eye,
* Patient presenting with chronic retinal pathologies other than AMD, defined according to the modified international AREDS study (Ferris et al. 2013) , in the included eye,
* Patient taking systemic drugs with an immunomodulatory action: immunosuppressants, immunomodulators, chemotherapy or corticosteroids,
* Patient with systemic pathologies modifying their immune status,
* Patient with a history of diabetes,
* Patient who had dynamic phototherapy on the included eye.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of the survival of human monocytes on ARPE-19 cultures, between the group of patients with atrophic AMD and patient with no retinal pathology (control). | through study completion, an average of 1 year
  Survival will be evaluated by automated counting of monocytes

SECONDARY OUTCOMES:
Comparison of human monocyte survival on ARPE-19 cell lines between different groups of patients with AMD or according to severity of disease. | through study completion, an average of 1 year
  Survival will be assessed by automated counting of monocytes on the culture plate after specific immunostaining of the monocytes.
Comparison of alterations in ARPE-19 cells lines after culture by human monocytes: | through study completion, an average of 1 year
  Comparison of alterations in ARPE-19 cells lines after culture by human monocytes:
  * Between the atrophic AMD group and the control group,
  * With respect to the stage of the AMD (early / intermediate AMD, exudative or atrophic AMD),
  * With respect to the evolving profile of atrophic AMD defined by autofluorescence examination,
  * With respect to the severity of the clinical involvement of atrophic AMD,
  * With respect to the recognized risk factors of the disease (age, sex, smoking status and obesity).
  The alteration of ARPE-19 cells on expression level of OTX2, a ubiquitous transcription factor in EPR cells, will be studied. OTX2 is normally under-expressed in-vitro when a supernatant of lipopolysaccharide-activated monocytes is added to the culture medium.
To compare the secretion of IL1 from patient's monocytes: | through study completion, an average of 1 year
  To compare the secretion of IL1 from patient's monocytes:
  * Between the atrophic AMD group and the control group, With respect to the stage of the AMD (early / intermediate AMD, exudative or atrophic AMD),
  * With respect to the evolving profile of atrophic AMD defined by autofluorescence examination,
  * With respect to the severity of the clinical involvement of atrophic AMD,
  * With respect to the recognized risk factors of the disease (age, sex, smoking status and obesity).
  The secretory activity of monocytes on the following cytokines will be evaluated : IL1, IL6 and TNF by two techniques: qPCR and ELISA.
To compare the secretion of IL6 from patient's monocytes: | through study completion, an average of 1 year
  To compare the secretion of IL6 from patient's monocytes:
To compare the secretion of TNF from patient's monocytes | through study completion, an average of 1 year
  To compare the secretion of TNF from patient's monocytes:

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Mathis, MD, Principal Investigator — Service d'Ophtalmologie Hospices Civils de Lyon Hôpital de la Croix Rousse
Locations (2):
- France (2):
  - Hôpital Edouard Herriot, Lyon
  - Service d'ophtalmologie-HOSPICES CIVILS DE LYON - Hôpital de la Croix-Rousse, Lyon

IPD SHARING:
Plan to Share IPD: Undecided